CLINICAL TRIAL: NCT00958581
Title: A Prospective, Randomized, Double-blinded Single-site Control Study Comparing Blood Loss Prevention of Tranexamic Acid (TXA) to Epsilon Aminocaproic Acid (EACA) for Corrective Spinal Surgery
Brief Title: Tranexamic Acid (TXA) Versus Epsilon Aminocaproic Acid (EACA) Versus Placebo for Spine Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 08-779
Record Dates: First submitted 2009-08-11; First posted 2009-08-13 (Estimated); Results first posted 2017-12-12 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2017-12

CONDITIONS: Scoliosis
Keywords: antifibrinolytics
MeSH Terms: conditions — Scoliosis | interventions — Tranexamic Acid; Saline Solution; Aminocaproic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Normal Saline (Placebo Comparator): Patients infused with normal saline before and during the surgical procedure as a placebo.
  Interventions: Drug: Normal Saline
- Tranexamic acid (Experimental): Patients receive TXA before and during the surgical case.
  Interventions: Drug: Tranexamic Acid
- Epsilon Aminocaproic Acid (Experimental): Patients will receive EACA before and during the surgical case.
  Interventions: Drug: Epsilon aminocaproic acid

INTERVENTIONS:
Drug: Tranexamic Acid — For TXA, the loading dose is 10mg/kg infused over 15 minutes, while the maintenance dose is 1/mg/kg hr.
  Other Names: TXA
  Arms: Tranexamic acid
Drug: Normal Saline — Normal saline of same volume as the intervention group will be given as the intervention group as a loading dose and maintenance dose.
  Other Names: Placebo
  Arms: Normal Saline
Drug: Epsilon aminocaproic acid — For EACA, the loading dose is 100mg/kg infused over 15 minutes, while the maintenance dose is 10mg/kg hr.
  Other Names: Amicar, EACA
  Arms: Epsilon Aminocaproic Acid

SUMMARY:
Tranexamic acid (TXA) and epsilon aminocaproic acid (EACA) have been reported to reduce blood loss in the cardiac surgery literature but they have not been reported in use head-to-head in the orthopedic surgery literature. In a randomized, double-blind, prospective study we believe that TXA will be more effective than both EACA and placebo at reducing blood loss for corrective spinal surgery.

DETAILED DESCRIPTION:
Study Design The study is designed as a prospective, randomized, double-blinded control trial. The patient, researcher, surgeon, and anesthesiologist will all be blinded to the patient's treatment. Patients will either receive TXA, EACA, or normal saline. The study will determine and compare differences in blood loss intra-operatively and estimate blood loss postoperatively through monitoring of subfascial Hemovac drain outputs at the incision site between the three groups. Postoperatively, laboratory values, drain outputs, and clinical outcomes will be carefully followed.

The primary goal of this study is to compare the efficacy of TXA to EACA to placebo in patients undergoing corrective spinal surgery for adolescent idiopathic scoliosis (AIS), neuromuscular scoliosis (NMS), and with adult deformity (AD). Outcome measures will include intra-operative and perioperative blood loss, transfusion rates, complete blood counts, and coagulation profiles, as well as postoperative wound drainage, complications, and length of stay.

Standardized treatment protocol For EACA, the loading dose is 100mg/kg infused over 15 minutes, while the maintenance dose is 10mg/kg hr. For TXA, the loading dose is 10mg/kg infused over 15 minutes, while the maintenance dose is 1/mg/kg hr. Since TXA is prepared by pharmacy at a concentration ten times less than the concentration of EACA, the volume of medication administered during the loading and maintenance phase is identical. This is the ideal method for physician blinding and has been discussed in depth with the anesthesia department. The dosing regimen is also in accordance with existing guidelines and current literature. The literature also reports safely using TXA at a 100mg/kg loading dose followed by a 10mg/kg hr maintenance dose. However, improved efficacy at this higher dose of TXA has not been proven in a single orthopedic study. Since TXA is reported to be ten times more potent than EACA, delivering a dose of TXA that is ten times smaller than EACA is valid and well supported in the literature.

Surgical correction of the spine Dorsal lumbar access is achieved by a posterior lumbar skin incision along the midline. Paravertebral muscles are dissected away from bony structures taking care to achieve adequate hemostasis. Multi-level spinal osteotomies and/or releases of bony and ligamentous structures are performed to increase mobility of the spinal column. Bone grafts consisting of autologous bone or allograft are filled in to allow for bony fusion of the spinal column and limit motion. Pedicle screws are placed segmentally into vertebral bodies to provide adequate fixation of rod instrumentation. Stainless steel, titanium, or cobalt rods are placed to help correct and stabilize the spine while fusion occurs. Generally the greatest blood loss occurs during dissection and placement of pedicle screws while rod placement is associated with less blood loss. Subfascial Hemovac or Jackson-Pratt drains are placed at the wound site during closure to allow for adequate drainage and determination of post-operative blood loss.

Investigation schedule and follow-up Data will be collected pre-operatively regarding individual patient demographics, laboratory values, and the surgical procedure to be performed. Intra-operatively, data will be gathered to estimate blood loss and account for changes in fluid balance. Anesthesiologists are asked to maintain a MAP of 60 during the surgical exposure and anchor placement and a MAP of 70-90 during the surgical correction. Similarly, surgeons are asked to place only subfascial Hemovac drains at the incision site. These are both standard practice and have . Postoperatively, laboratory values, drain output, and clinical outcomes are carefully followed until the patient is discharged. Given the increased risk of renal failure with the use of Aprotinin changes in BUN to CR ratio are carefully monitored post-operatively. This data is recorded onto a de-identified data collection sheet by the researchers. These patient data sheets are then entered onto a protected electronic database, while the data sheets are stored as a back-up until the study is complete. Once the completed database is analyzed and summarized, the results will be presented to the involved participants without any identifiable patient information.

Statistical considerations While useful, this analysis is limited by the great variability in study design and control groups between prior orthopedic studies. Since no orthopedic study has compared TXA and EACA together, conducting a power analysis required pooling of data from two or three studies. This proved difficult, as control groups were dissimilar between the studies.

Power analysis was performed multiple times using data from several studies. When estimating the sample size required comparing TXA and EACA, attempts were made to choose two studies with similar intra-operative blood losses within the control groups. A cardiac study, albeit with dissimilar sample variance, was also used to estimate the sample size needed for this study. Finally, determining the sample size for outcomes of total blood loss and transfusion requirements proved difficult as even fewer studies reported these outcomes. Blood loss will be estimated in the operation room, but will also be calculated taking into account patient body mass, pre/postoperative hematocrit, and relative fluid balance. This will minimize the variance in reported blood loss. A power analysis will be performed again once 60 patients with AIS, NMS, or AD have been enrolled into the study.

With a single institution of surgeons and anesthesiologists participating in the study, we expect a smaller variation in operative blood loss than reported in prior studies. Data will not only be analyzed for all patients collectively, but will also be stratified by diagnosis (AIS, NMS, and AD). The purpose of stratifying into these groups is threefold. First, separation by diagnosis allows for more diligent control of patient-related factors that may affect blood loss and transfusion rate. Secondarily, stratification by diagnosis allows for a better understanding of which patients benefit most from one treatment option over another. Lastly, it allows for a broader application of the results from this study not only to patients with AIS, but to all spinal deformity patients.

An analysis of variance, univariate, and multivariate logistic regression analysis will be used to analyze the difference in outcomes. Odds ratios will be calculated regarding the risk for autologous or allogenic transfusion both intra and postoperatively. P-values will be calculated regarding the relative blood loss in the intra and postoperative periods as well. The groups will be analyzed to characterize the homogeneity of their pre-operative characteristics that may influence blood loss. Patients with AIS, NMS or AD will be stratified by primary diagnosis and analyzed separately but also collectively accounting for patient and surgery-related confounders. Non-continuous data will be analyzed with a non-parametric test. Pre-operative curve characteristics including Cobb angle and number of vertebrae fused will be categorized to ensure similar groups for comparison.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing thoracic and/or lumbar surgery for correction of adolescent idiopathic scoliosis, neuromuscular scoliosis, or adult deformity for correction of condition via posterior spinal fusion of 6 levels or greater.

Exclusion Criteria:

* No renal dysfunction identified by elevated blood urea nitrogen (BUN) and creatinine (CR) or BUN to CR ratio greater than 20:1
* Hold religious and/or other beliefs limiting blood transfusion
* Currently use anti-coagulant medication or have past medical history leading to abnormal coagulation profile pre-operatively
* Significant past medical history preventing the use of TXA or EACA described in the protocol

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2008-12; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J Errico, MD, Principal Investigator — New York University School of Medicine - Department of Orthopaedic Surgery; Baron S Lonner, MD, Principal Investigator — New York University - Department of Orthopaedic Surgery
Locations (1):
- New York University School of Medicine - Department of Orthopaedic Surgery - Spine, New York, New York, United States

REFERENCES:
- [Derived] Verma K, Errico TJ, Vaz KM, Lonner BS. A prospective, randomized, double-blinded single-site control study comparing blood loss prevention of tranexamic acid (TXA) to epsilon aminocaproic acid (EACA) for corrective spinal surgery. BMC Surg. 2010 Apr 6;10:13. doi: 10.1186/1471-2482-10-13. PMID 20370916
- See also: BMC Surgery, April 2010 — http://link.springer.com/article/10.1186%2F1471-2482-10-13

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Consenting completed at PI and co-investigators' private offices, clinic and in preoperative center. Study staff approved by the IRB consent the patients. First patient enrolled on 12/16/2008. Last patient enrolled on 9/17/2012.
Pre-assignment Details: Patients were excluded from the trial after enrollment if their surgery was cancelled.
Groups:
- Epsilon Aminocaproic Acid: Patients will receive EACA before and during the surgical case.
  Epsilon aminocaproic acid : For EACA, the loading dose is 100mg/kg infused over 15 minutes, while the maintenance dose is 10mg/kg hr.
- Normal Saline: Patients infused with normal saline before and during the surgical procedure as a placebo.
  Normal Saline :
- Tranexamic Acid: Patients receive TXA before and during the surgical case.
  Tranexamic Acid : For TXA, the loading dose is 10mg/kg infused over 15 minutes, while the maintenance dose is 1/mg/kg hr.
Period: Overall Study
Arm/Group | Epsilon Aminocaproic Acid | Normal Saline | Tranexamic Acid
Started | 61 | 61 | 55
Completed | 61 | 61 | 55
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Epsilon Aminocaproic Acid | Normal Saline | Tranexamic Acid | Total
Number analyzed (Participants) | 61 | 61 | 55 | 177
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 42 | 47 | 36 | 125
  Between 18 and 65 years | 15 | 12 | 11 | 38
  >=65 years | 4 | 2 | 8 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 39 | 45 | 134
  Male | 11 | 22 | 10 | 43
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 61 | 61 | 55 | 177

OUTCOME MEASURES:

1. Primary Outcome: Total Blood Loss Over Course of Stay (Intraoperative and Postoperatively Until Discharge)
Time Frame: 1 Week
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Epsilon Aminocaproic Acid | Normal Saline | Tranexamic Acid
Number analyzed (Participants) | 61 | 61 | 55
ml | 1775 (853) | 2116 (1201) | 1531 (911)

2. Secondary Outcome: Total Units of Autologous and Allogenic Transfusion (Both Intraoperatively and Postoperatively Until Discharge)
Time Frame: 1 week
Population: Data for this outcome measure unattainable as PI and study team are no longer with the institution. This outcome measure data was not published in paper.
Arm/Group | Normal Saline | Tranexamic Acid | Epsilon Aminocaproic Acid
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Length of Hospital Stay From Admission Until Patient Discharge
Time Frame: 1 week
Population: as for outcome 2
Arm/Group | Normal Saline | Tranexamic Acid | Epsilon Aminocaproic Acid
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Epsilon Aminocaproic Acid | Normal Saline | Tranexamic Acid
Serious Adverse Events (participants affected / at risk) | 1/61 | 1/61 | 1/55
Other Adverse Events (participants affected / at risk) | 0/61 | 0/61 | 0/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Epsilon Aminocaproic Acid (N=61) | Normal Saline (N=61) | Tranexamic Acid (N=55)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No